CLINICAL TRIAL: NCT01163084
Title: A Randomized Phase Ib/II Study of Preoperative GDC-0449 and Androgen Ablation Compared to Androgen Ablation Alone Followed by Radical Prostatectomy for Select Patients With Locally Advanced Adenocarcinoma of the Prostate
Brief Title: Leuprolide Acetate or Goserelin Acetate With or Without Vismodegib Followed by Surgery in Treating Patients With Locally Advanced Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-01737; NCI-2010-01737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000670590; 2009-0473 (Other: M D Anderson Cancer Center); 8384 (Other: CTEP); N01CM00039 (NIH); N01CM62202 (NIH); P30CA016672 (NIH); U01CA062461 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Prostate Adenocarcinoma; Stage IIA Prostate Cancer AJCC v7; Stage IIB Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Leuprolide; luprolide acetate gel depot; HhAntag691

ARMS (2):
- Arm I (leuprolide acetate, goserelin acetate, vismodegib) (Experimental): Patients receive LHRH analogue comprising leuprolide acetate IM or goserelin acetate SC on day 1 and vismodegib PO QD on days 1-28. Treatment repeats every 28 days for up to 16 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Drug: Vismodegib
- Arm II (leuprolide acetate, goserelin acetate) (Active Comparator): Patients receive LHRH analogue comprising leuprolide acetate or goserelin acetate as in Arm I. Treatment repeats every 28 days for up to 16 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Goserelin Acetate; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (leuprolide acetate, goserelin acetate, vismodegib)
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
  Arms: Arm I (leuprolide acetate, goserelin acetate, vismodegib)

SUMMARY:
This randomized phase I/II trial studies giving leuprolide acetate or goserelin acetate together with or without vismodegib followed by surgery to see how well they work in treating patients with prostate cancer that has spread from where it started to nearby tissue or lymph nodes. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide acetate or goserelin acetate, may lessen the amount of androgens made by the body. Vismodegib may slow the growth of tumor cells. Giving antihormone therapy together with vismodegib may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the difference in less than or equal to 5% tumor involvement between patients between the two arms.

SECONDARY OBJECTIVES:

I. To assess differences in hedgehog signaling, androgen signaling, markers linked to high grade prostate cancer (PCa) progression, proliferation, apoptosis, and the expression of androgen producing enzymes in the tumor microenvironment between the two arms.

II. To assess safety of preoperative GDC-0449 (vismodegib) in combination with luteinizing hormone-releasing hormone (LHRH).

III. To assess the difference in proportion of patients with negative disease surgical margins between the two arms.

IV. To collect and archive tissue from the primary tumor, bone marrow and blood (serum, plasma), bone marrow aspirate for future study.

V. To assess difference in relapse rate (biochemical, objective) and time to progression.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (androgen-ablation therapy and vismodegib): Patients receive LHRH analogue comprising leuprolide acetate intramuscularly (IM) or goserelin acetate subcutaneously (SC) on day 1 and vismodegib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 16 weeks in the absence of disease progression or unacceptable toxicity.

ARM II (androgen-ablation therapy): Patients receive LHRH analogue comprising leuprolide acetate or goserelin acetate as in Arm I. Treatment repeats every 28 days for up to 16 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients undergo radical prostatectomy.

After completion of study therapy, patients are followed up every 6 months for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of prostatic adenocarcinoma via a minimum of 6 core biopsy samples
* Clinical stage T1c or T2 with high-grade disease (Gleason's 8-10) on initial biopsy and prostate specific antigen (PSA) > 10 ng/ml, or clinical stage T2b-T2c with Gleason's grade >= 7
* No evidence of metastatic disease as determined by imaging
* Initial therapy with antiandrogen treatment is allowed but must be within 4 weeks prior to study enrollment
* Appropriate surgical candidate for radical prostatectomy and an Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absence of major co-morbidity as determined by the treating physician
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >=100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have prothrombin time (PT), partial thromboplastin time (PTT) and fibrinogen levels within institutional normal limits and no history of substantial non-iatrogenic bleeding diathesis
* Men and their female partners must agree to use two forms of contraception (i.e., barrier contraception and one other method of contraception) during study treatment and for at least 12 months post-treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Histologic variants in the primary tumor (histologic variants other than adenocarcinoma)
* Patients who have had chemotherapy or radiotherapy for prostate cancer prior to entering the study
* Patients who have received prior treatment with GDC-0449
* Patients may not be receiving any other investigational agents
* Patients receiving previous androgen ablation or current androgen ablation of greater than 4 week's duration
* Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing causes of death (such as but not limited to, unstable angina, myocardial infarction within the previous 6 months, or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia, uncontrolled hypertension)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or LHRH analogues
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically important (in the opinion of the treating physician) history of liver disease, including viral or other hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with prior malignancy if there is an increased chance (>= 30%) of relapse in the following five years (in the opinion of the treating physician)
* Patients who have received systemic treatment for cancer within the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Karlou M, Tzelepi V, Efstathiou E. Therapeutic targeting of the prostate cancer microenvironment. Nat Rev Urol. 2010 Sep;7(9):494-509. doi: 10.1038/nrurol.2010.134. PMID 20818327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by physicians in the Genitourinary Medical Oncology Clinic and Urology clinic.
Pre-assignment Details: 10 participants started but only 9 were randomized
Groups:
- Group A- GDC-0449 and Androgen Ablation (LHRHa): Group A will receive 150mg GDC-0449 daily for 3 months prior to radical prostatectomy.
- Group B- Androgren Ablation (LHRHa) Alone: Patients will receive an LHRHa (monthly injection or three-month injection) for a maximum of 4 months before a prostatectomy is performed.
Period: Overall Study
Arm/Group | Group A- GDC-0449 and Androgen Ablation (LHRHa) | Group B- Androgren Ablation (LHRHa) Alone
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group- B Androgren Ablation (LHRHa) Alone: Patients will receive an LHRHa (monthly injection or three-month injection) for a maximum of 4 months before a prostatectomy is performed.
- Total: Total of all reporting groups
Arm/Group | Group A- GDC-0449 and Androgen Ablation (LHRHa) | Group- B Androgren Ablation (LHRHa) Alone | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 63 [55 to 72] | 63 [62 to 66] | 63 [55 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With =< 5% Tumor Involvement
Description: Each patient's pathologic staging will be assessed from the samples collected from prostatectomy. Will be descriptively summarized. Two-sided Chi-Square test will be used to provide the test of significance between the 2 groups of LHRHa versus LHRHa plus vismodegib.
Time Frame: Baseline up to 4 months or radical prostatectomy, whichever comes first
Population: Results was not determined.
Groups:
- Group A-GDC-0449 and Androgen Ablation (LHRHa: Group A will receive 150mg GDC-0449 daily for 3 months prior to radical prostatectomy
- Group B Androgen Ablation (LHRHa) Alone: Patients will receive an LHRHa (monthly injection or three-month injection) for a maximum of 4 months before a prostatectomy is performed.
Arm/Group | Group A-GDC-0449 and Androgen Ablation (LHRHa | Group B Androgen Ablation (LHRHa) Alone
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Differences in Relapse Rates by PSA Levels (Biochemical)
Description: Will be descriptively summarized.
Time Frame: Date of surgery, then every 6 months, up to 8 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Time to PSA (Biochemical) Progression, Defined as PSA Recurrence
Description: Will be descriptively summarized. PSA recurrence is defined as two (2) serial measureable rises in PSA concentration above the undetectable level with the standard assay (> 0.1 ng/mL).
Time Frame: From the date of surgery and elevated post operative PSA concentration, assessed up to 8 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Time to PSA (Clinical) Progression, Defined as a Serial Rise in PSA Concentration in the Presence of Castrate Serum Testosterone Concentration or Radiographic Evidence of Progression
Description: as for outcome 3
Time Frame: From the date of surgery and elevated post operative PSA concentration, assessed up to 8 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Proportion of Patients With PSA =< 0.2 ng/mL
Description: Will be descriptively summarized.
Time Frame: Up to 8 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Differences in the Rate of Positive Surgical Margins Between the Two Groups
Description: Will be descriptively summarized.
Time Frame: Baseline to up to 8 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Differences in Relapse Rates by Bone Scan/Computed Tomography Scan (Objective)
Description: Will be descriptively summarized.
Time Frame: Baseline to up to 8 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Proportion of Patients Expressing Differences in Hedgehog, Androgen Signaling and Related Genes Markers
Time Frame: Up to 8 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During on-study tests/visits that occur every 4 weeks for all participants until the follow up visit after radical prostatectomy, assessed up to 5 months.
Description: All adverse events reported as routine part of a clinical trial.
Arm/Group | Group A- GDC-0449 and Androgen Ablation (LHRHa) | Group B- Androgren Ablation (LHRHa) Alone
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A- GDC-0449 and Androgen Ablation (LHRHa) (N=4) | Group B- Androgren Ablation (LHRHa) Alone (N=5)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholesterol, high (Investigations) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Edema Limbs (Blood and lymphatic system disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
Headache (Nervous system disorders) | 1 | 0
Hot flashes (Vascular disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 4
hypotension (Vascular disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pustular (Skin and subcutaneous tissue disorders) | 0 | 1
Spasticity (Nervous system disorders) | 1 | 0
Urinal frequency (Renal and urinary disorders) | 0 | 1
Watering eyes (Eye disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less